CLINICAL TRIAL: NCT06247618
Title: Virtual Reality as a Tool to Promote Healthcare Providers Wellbeing in Pediatric Palliative Care
Brief Title: Virtual Reality for Pediatric Palliative Care Team
Acronym: PPCVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Anna Marinetto, RN, RN, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ppcVirtualReality
Record Dates: First submitted 2023-09-07; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Occupational Stress
Keywords: virtual reality; pediatric palliative care; anxiety; burnout
MeSH Terms: conditions — Occupational Stress; Anxiety Disorders; Burnout, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (Experimental)
  Interventions: Device: visor

INTERVENTIONS:
Device: visor — The treatment will have a duration of 4 weeks, with the execution of two sessions per week with the use of a viewer positioned on the head that allows users to navigate and interact in real time with a three-dimensional (3D) environment

SUMMARY:
Is virtual reality a useful and usable tool to improve the psychological well-being of PPC operators? study primary obtv: assessment of occupational psychological well-being (divided into stress, depression, anxiety and risk of burnout) in the population of health professionals working in pediatric palliative care; verify if the virtual reality tool leads to an improvement change at the level of the investigated items (feasibility study). The treatment will have a duration of 4 weeks, with the execution of two sessions per week with the use of a viewer positioned on the head that allows users to navigate and interact in real time with a three-dimensional (3D) environment At time zero (T0), the participants will be administered, shortly before the application of virtual reality, the Mini-Z survey 2.0 questionnaires (the single item burnout question), Depression Anxiety Stress Scales 21 (DASS-21), and a demographic questionnaire (gender, age, profession, shift work, years of work in PPCs). At the end of the compilation, two vision treatments will follow, which will take place three to four days apart.

At time T1 (second week) and time T2 (third week) the DASS-21 will initially be administered followed by two weekly treatments with a visor. At the end (T3) the compilation of both tests (Mini-Z survey 2.0-the single item burnout question and the DASS-21) will be repeated following the last two applications of the viewer.

ELIGIBILITY:
Inclusion Criteria:

* work within the pediatric hospice of Padua
* Absence of neurological pathologies
* personnel who actively engage in membership/participation during all 4 weeks of the project

Exclusion Criteria:

* Subject do not sign written consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
the psychological well-being of healthcare providers: risk of burnout | Data collection lasted for four weeks
  - Mini-Z Survey 2.0 (single-item): examines the risk of burnout among healthcare provides, particularly The Mini-Z responds to the goal of framing/identifying the burnout risk of workers on the pediatric palliative care team. , it was analysed frequencies and percentages of burnout risk based on the analysis criteria identifiable in Nagasaki et al. 2022 (1- "In Total burnout"; 2-"Always has burnout symptoms the burnout symptoms I perceive are persistent"; 3-"Beginning of burnout"; 4-"Under stress"; 5-"Never felt in Burnout").
the psychological well-being of healthcare providers: anxiety, depression and stress | Data collection lasted for four weeks
  - DASS-21(the Depression Anxiety Stress Scales 21) DASS-21 is a psychometric self-assessment test, derived from the Depression Anxiety Stress Scales [22], detecting three constructs: anxiety, depression and stress. It is measured by 21 items on a 4-point Likert scale (from "0-Not at all applies to me" to "3-It applies a lot or most of the time to me"). Cronbach's alpha of .80 is very good evidence of the high reliability of the tool's content.

CONTACTS AND LOCATIONS:
Overall Officials: Zanin, Principal Investigator — Azienda Ospedale-Università Padova
Locations (1):
- Hospice Pediatrico- Azienda Ospedale Università Padova, Padua, PD, Italy